CLINICAL TRIAL: NCT07406893
Title: Reduction of Bacterial Seeding in Total Shoulder Arthroplasty: Prontosan Antimicrobial Gel Incision Preparation Versus No Preparation in Male Patients
Brief Title: Reduction of Bacterial Seeding in Total Shoulder Arthroplasty
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: St. Louis University (Other)
Collaborators: Innovice, LLC (Unknown); American Shoulder and Elbow Surgeons (Other)
Responsible Party: Principal Investigator, Randall J. Otto, MD, Associate Professor, St. Louis University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Study00000436
Record Dates: First submitted 2026-02-05; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Joint Arthroplasty; Shoulder; Cutibacterium Acnes; Prosthetic Joint Infection
Keywords: Antimicrobial wound gel; Dermal layer; Skin preparation

STUDY DESIGN:
Intervention Model Description: This is a prospective clinical trial in which patients will be assigned a study arm in sequential fashion.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- No skin incision preparation (No Intervention): All patients will receive standard pre-operative prophylactic antibiotics and external skin preparation prior to draping. At the time of the surgery, after the skin incision has been made with a skin knife, the dermal layer will not be prepped with any additional agents for patients in this arm.
- Prontosan Wound Gel (Experimental): All patients will receive standard pre-operative prophylactic antibiotics and external skin preparation prior to draping. At the time of the surgery, after the skin incision has been made with a skin knife, the dermal layer will be prepped with Prontosan Wound Gel for patients in this arm. Prontosan Wound gel is an antimicrobial gel agent intended to keep wounds free of bacteria.
  Interventions: Device: Prontosan Wound Gel

INTERVENTIONS:
Device: Prontosan Wound Gel — Applied to dermal layer of skin after incision is made for surgery.
  Arms: Prontosan Wound Gel

SUMMARY:
The purpose of this study is to compare the growth of intra-operative tissue cultures of Cutibacterium Acnes after primary shoulder replacement when using a no-prep control group versus Prontosan wound gel applied to the skin layer after the skin incision has been made.

DETAILED DESCRIPTION:
60 male patients undergoing primary anatomic or reverse shoulder arthroplasty will be enrolled in this prospective, randomized controlled trial evaluating the use of Prontosan wound gel versus no preparation to the dermal layer of skin after incision has been made. Participants will be randomly assigned to one of two groups of 30 patients: control (no post-incision dermal preparation) and Prontosan antimicrobial gel application to the dermal layer after skin incision. All patients, regardless of assignment, receive the same pre-incision skin preparations, prophylactic antibiotics, and intraoperative irrigation. After final implantation and before wound closure, culture swabs will be obtained (2 deep cultures, 2 superficial, and 1 implant). All cultures will be held in the lab for 2 weeks to monitor for growth of C. acnes.

ELIGIBILITY:
Inclusion Criteria:

* Adult male 18 years of age or older undergoing elective primary total shoulder arthroplasty, including both anatomic and reverse total shoulder arthroplasty, for indications including massive rotator cuffs, rotator cuff arthropathy, glenohumeral osteoarthritis, and acute fractures.

Exclusion Criteria:

* Any revision shoulder arthroplasty procedure or other shoulder surgery that is not a primary shoulder arthroplasty.
* Patients with allergy to active ingredients in Prontosan gel
* Patient is unable to consent for themselves
* Patient is non-English speaking
* Females

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Presence of bacteria within shoulder cultures | 14 days
  Each participant will have culture swabs taken at the end of the surgical case from deep, superficial, and implant locations. Cultures will be held in the lab for 2 weeks to evaluate for the presence of bacteria.

CONTACTS AND LOCATIONS:
Overall Officials: Randall Otto, MD, Principal Investigator — St. Louis University
Locations (1):
- Saint Louis University, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No